CLINICAL TRIAL: NCT06206590
Title: Analysis of Differential Proteins and Maternal Influencing Factors of Septic Shock in Neonates Born to ≤32-week Preterm Infants or Infected Mothers During Pregnancy
Brief Title: Analysis of Differential Proteins and Maternal Influencing Factors of Septic Shock in Neonates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, Ma Dongju, Physician, Guangdong Women and Children Hospital
Other Study IDs: 202301393
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Neonatal Disease
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exposed group: Contains differential proteins
  Interventions: Other: Whole-proteomic assay
- non-exposed group: No differential protein
  Interventions: Other: Whole-proteomic assay

INTERVENTIONS:
Other: Whole-proteomic assay — Whole-proteomic analysis was performed on all the blood samples

SUMMARY:
1. Explore 32 weeks of premature infants or maternal pregnancy infection of newborn septic shock maternal influence factors. 2. Through maternal blood samples before delivery and labor cord blood sample screening and septic shock related proteomics analysis, explore the relationship between the difference protein and septic shock and prognosis, and explore the pathway mechanism, in order to prevent and reduce the occurrence of septic shock in premature infants

DETAILED DESCRIPTION:
The birth cohort was established with 32 weeks of premature infants or maternal infection during pregnancy.Whole proteomic analysis was performed on maternal blood before delivery and umbilical cord blood samples at delivery,and screscreen differential proteins associated with septic shock and classify these proteins as leak factor into exposed and non-exposed groups for cohort study.The incidence and mortality of shock,severe brain injury and BPD in the two groups were compared, and the mechanism of the differential protein was studied to provide early warning in children with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* All ≤32-week premature infants admitted to our NICU; All newborns delivered by the mother infected during pregnancy

Exclusion Criteria:

* Not delivered in our hospital; congenital cardiovascular development malformation, fetal malformation, genetic metabolic diseases, etc

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns who born in Guangdong Women and Children Hospital
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and mortality of shock | 1/10/2025

CONTACTS AND LOCATIONS:
Overall Officials: xiuzhen ye, Study Chair — Guangdong Women and Children Hospital
Locations (1):
- Guangdong Women and Children Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
after the end of the study